CLINICAL TRIAL: NCT06836635
Title: Comparative Study Between Ultrasound-Guided Erector Spinae Plane Block and Thoracic Paravertebral Block for Postoperative Analgesia After Video-Assisted Thoracoscopic Surgery
Brief Title: Postoperative Analgesia After Video-Assisted Thoracoscopic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: FMASU MS99/2024
Record Dates: First submitted 2025-01-05; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2024-03

CONDITIONS: Postoperative Pain Management, After VATS
Keywords: Postoperative pain management

STUDY DESIGN:
Intervention Model Description: Post operative pain control
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The ESPB group (Experimental): a high-frequency linear ultrasound probe will be placed in a longitudinal orientation 3 cm from the midline. Once the erector spinae muscle and the transverse processes identified, a 100mm needle (B- Braun Medical Inc., Bethlehem, PA, USA) will be inserted after standard skin disinfection in a caudad-to-cephalad direction using a sterile probe cover until the tip lay in the interfacial plane deep to the erector spinae muscle. After hydrolocalization with normal saline, this plane will be opened. 20 milliliters (mL) of 0.25% bupivacaine will be administered for block performance.
  Interventions: Procedure: ESPB group
- The TPVB group (Experimental): A high-frequency linear ultrasound probe will be placed in a vertical orientation 23 cm lateral to the midline. Once the transverse process, internal intercostal membrane and parietal pleura identified, a 100mm needle (B- Braun Medical Inc., Bethlehem, PA, USA) will be inserted after standard skin disinfection laterally to medically Use a sterile probe cover until the tip lay in the thoracic paravertebral space beyond the internal intercostal membrane. After injection with normal saline, to confirm ventral pressing of the parietal pleura, 20 mL of 0.25% bupivacaine will be administered for block performance
  Interventions: Procedure: TPVB group

INTERVENTIONS:
Procedure: ESPB group — The patient will be placed in the lateral position. Block will be performed under complete aseptic precautions using ultrasound machine with high frequency linear probe covered with sterile sheath .
  The block will be performed at the T5-T6 level of the spine using an in-plane approach. Sensory block of the 5th intercostal space in the midaxillary line will be assessed by unilaterally using cold perception until 30 minutes after nerve block. If sensory blockade did not occur, the patient will be excluded from the study.
  Arms: The ESPB group
Procedure: TPVB group — The patient will be placed in the lateral position. Block will be performed under complete aseptic precautions using ultrasound machine with high frequency linear probe covered with sterile sheath .
  The block will be performed at the T5-T6 level of the spine using an in-plane approach. Sensory block of the 5th intercostal space in the midaxillary line will be assessed by unilaterally using cold perception until 30 minutes after nerve block. If sensory blockade did not occur, the patient will be excluded from the study.
  Arms: The TPVB group

SUMMARY:
Video-assisted thoracoscopic surgery (VATS) is a commonly performed minimally invasive procedure that has lead to lower levels of pain. However, VATS require analgesia that blocks both visceral and somatic nerve fibers for more effective pain control.

In this study investigators will compare the analgesic effect of ultrasound guided erector spinae plane block (ESPB) and thoracic paravertebral block (TPVB) after VATS.

DETAILED DESCRIPTION:
All patients will be assessed preoperatively by careful history taking, full physical examination, laboratory evaluation and other appropriate investigations.

At the preoperative visit, all patients will be instructed on how to evaluate their own pain by using a 10-cm visual analog pain scale (0= no pain, 10= maximum pain imaginable).

The nerve block will be performed in the preoperative block area following standardized monitoring, including noninvasive blood pressure (BP), electrocardiogram (ECG), and pulse oximetry (PO). Oxygen 23 L/min was applied through the nasal cannula, and midazolam 0.025 mg/kg iv, will be given.

All blocks will be performed by the same two experienced senior attending doctors in ultrasound-guided nerve blocks. Patients will be randomly assigned into one of the following groups using computer generated codes and closed opaque sealed envelopes and patient and anesthesiologist who collect data will not know which type of block administered (as block will be done in holding area):

Group 1 (TPVB group): patients will receive TPVB. Group 2 (ESPB group): patients will receive ESPB block. The patient will be placed in the lateral position. Both blocks will be performed under complete aseptic precautions using ultrasound machine with high frequency linear probe covered with sterile sheath .

The blocks will be performed unilateral at the T5-T6 level of the spine using an in-plane approach.

Pre-operative chest ultrasound will be done by the anesthesiologist to detect complications after the blockade (hematoma in the puncture site by direct visualization and pneumothorax by Barcode/Stratosphere sign).

ELIGIBILITY:
Inclusion Criteria:

* Age eligible >20 - <70 yrs.
* Sex eligible both sex.
* Patients with American Society of Anesthesiologists (ASA) physical status 13 who will be scheduled for VATS, with three trochar ports. The trochar ports will be made at the fifth and sixth to intercostal levels. The chest drain will be inserted before the skin closure at the seventh or eighth intercostal level.

Exclusion Criteria:

* ≤20 or ≥70 years old.
* Declining to give written informed consent.
* History of allergy to the medications used in the study.
* Contraindication to regional anesthesia (including coagulopathy (platelet count ≤ 80,000, INR ≥ 1.5) and local infection).
* hepatic impairment (INR ≥1.5, Bilirubin ≥2, Albumin ≤2).
* Renal dysfunction (GFR <50ml/min).
* Psychiatric disorder.
* Pregnancy.
* Body mass index (BMI) ≥40 or ≤18 kg/m2.
* VATS procedure converted to open.
* Patient with history of thoracic spine surgery.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-03-10 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2024-09-09 (Actual)

PRIMARY OUTCOMES:
To compare the post-operative morphine consumption in first 24 hours between ESPB and TPVB after VATS | From injection to 24 hours postoperative

SECONDARY OUTCOMES:
Post-operative pain severity assessed by visual analogue scale (VAS) (every 6 hr for 24 hr at rest and during cough). | From injection to 24 hours postoperative
Time of first request of rescue analgesia (rescue analgesia will be given in case of break through pain VAS ≥ 4 inform of 0.1mg/kg morphine). | From injection to 24 hours postoperative
Incidence of post-operative nausea and vomiting. | From injection to 24 hours postoperative
Incidence of complications (haematoma and pneumothorax). | From injection to 24 hours postoperative
Patient satisfaction during procedure (score 1-4 (1= very dissatisfied, 2= dissatisfied, 3= satisfied, 4= very satisfied)). | From injection to 24 hours postoperative
Patient satisfaction after 1st post-operative day (score 1-4 (1= very dissatisfied, 2= dissatisfied, 3= satisfied, 4= very satisfied)). | From injection to 24 hours postoperative
Procedure time from scanning to injection of local anesthetic (LA) correctly. | From injection to 24 hours postoperative
Anesthesiologist satisfaction about simplicity of block or fear from complications (score 1-4 (1= very dissatisfied, 2= dissatisfied, 3= satisfied, 4= very satisfied)) | From injection to 24 hours postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Toka R Mohamed, M.B.B.CH, Principal Investigator — Anesthesia resident at Ain shams university
Locations (1):
- Ain shams university, Cairo, Egypt, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All data will be shared
Supporting Information: Study Protocol, SAP, ICF
Access Criteria: Free